CLINICAL TRIAL: NCT05412485
Title: Does Increased Frequency of Robot-assisted Gait Training Improve Gait Functions and Quality of Gait in Children With Cerebral Palsy: A Single Blinded, Randomized Pilot Study
Brief Title: Gait Improvement After Increased Frequency of Robot-assisted Gait Training in Cerebral Palsy Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sharjah (Other)
Responsible Party: Principal Investigator, Meeyoung Kim, Assistant Professor, University of Sharjah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC-21-06-22-01-S
Record Dates: First submitted 2022-06-01; First posted 2022-06-09 (Actual); Last update posted 2022-06-09 (Actual); Status verified 2022-06

CONDITIONS: Cerebral Palsy Spastic Diplegia
Keywords: Randomized pilot study; Cerebral palsy; Robotic assisted gait training; gait function
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: A prospective single blinded parallet-group, randomized clinical trial would be conducted.
Who Masked: Outcomes Assessor
Masking Description: Outcome measure assessor will be blinded to the allocation. The child performance will be recorded and the score will be obtained by another assessor who is not aware about the date of the recorded video and not knowing of the allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): Lokomat Certified physiotherapists will perform robotic assisted gait trainings. It will be performed 4 times per a week with a duration of 30 minutes on the lokomat with a treatment of 6 weeks phase.
  Initially the Physical therapist will adjust the body -weight support at 70 % which will be gradually reduced until obtain flexion of the knees during stance phases. The lokomat certified physiotherapist will monitor the condition of the knees and adjust the body weight support during the training.
  The Gait speed will be set at 0.7 km/hour and will gradually increase according to the comfortable speed selected by the child. The gait speed, Body weight support and the guidance force of the Lokomat will be adjusted and modified individually according to the ability of the child.
  Virtual reality games will be used to motivate the participants and verbal encouragement will be used to increase their adherence to the intervention.
  Interventions: Other: Robotic assisted gait training
- Control group (Active Comparator): The same procedures will be given twice a week frequency.
  Interventions: Other: Robotic assisted gait training

INTERVENTIONS:
Other: Robotic assisted gait training — Robotic assisted gait training is advanced technology used in the rehabilitation of neurological injuries and conditions like spinal cord injury, brain injury, stroke, multiple sclerosis, Parkinson's, cerebral palsy. It provides a repetitive task-specific motor training and modulates afferent input to spinal cord to generate rhythmic gait patterns that may be transformed to overground walking. The intensive repetitions of the rhythmic stepping movement during the training stimulates dependent plasticity and it may lead to brain reorganization. It facilitates cortical neural activities associated with motor control of walking.

SUMMARY:
Robot-assisted gait training (RAGT) can provide a longer training duration with a higher repetition of stepping while maintaining a stable pattern of movement. However, the existing evidence of its effectiveness is not clear. The aim of this study is to investigate the feasibility and the effect of increased frequency (4 times per week) of RAGT compared to the most common frequency (2 times per week). we hypothesize that increased frequency of RAGT will result in greater improvements on the gait functions. This research will investigate the effect of increased frequency on robotic assisted gait training (RAGT) in a frequency of 4 times per a week, and will compare the effect of robotic assisted gait training (RAGT) with increased frequency and with usual frequency (2 times per a week) in regards with gait functional parameters such as balance, speed, endurance, and quality of gait among cerebral palsy (CP) children's.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is defined as a group of disorders that affect mobility and posture with heterogeneous impairments such as muscle tone alternation, reduced selective motor control, joint contracture, postural control impairment and weakness of muscles. Independent walking is a priority goal for a lot of parents and children with CP.

RAGT has been considered as a revolutionary technology for gait enhancement. Lokomat, as one of RAGT devices, provides the intensive gait training with a number of repetitions of stepping while it preserves consistent pattern of movement. Lokomat with additional virtual reality games adds fun and challenge and enhances the involvement and motivation throughout the whole session. We will use Lokomat for RAGT for 6 weeks phase for both treatement and control groups. Only difference between groups is the frequency: 4 times a week for treatment group and 2 times a week for intervention group.

General gait and standing function will be measured by Gross motor function measure dimension E and D. Speed, endurance, balance, and quality of gait would be measured by 10 meter walk test, 6 minutes walk test, pediatric balance scale, and Edinburgh visual gait score. To our knowledge no previous studies investigated the effect of the increased frequency in RAGT with lokomat on improving gait speed, endurance, balance and quality in children with CP.

ELIGIBILITY:
Inclusion Criteria:

* children with spastic diplegia; being able to walk independently with or without using walking aids on at least 10 meters; classified as level Ι, II and ΙΙΙ in the gross motor function classification system (GMFCS).
* Children who can follow instructions of gross motor function measure (GMFM) testing and able to express discomfort and pain by verbal or nonverbal signs, having required range for lokomat (hip and knee flexion contracture ≤10°, knee valgus ≤40°, femur length ≥ 23 cm).

Exclusion Criteria:

* If they received botulinum toxin injections or underwent surgical intervention at least a year before the 6-week of the intervention or participated in another Lokomat training regime within the last 3 months.
* If they have: (a) fixed contractures and/or with bone instability; (b) seizure disorder that is not controlled by medication (if on medication, must not have had a seizure in the last 12 months); (c) baclofen infusion pumps in situ, open skin lesions and vascular disorder of lower extremities.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2022-06-07 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-07-30 (Estimated)

PRIMARY OUTCOMES:
The change in Gross motor function measure - Dimension E (GMFM E) between pre-treatment and post-treatment | will be measured at two intervals; pre-treatment and immediately after treatment
  it evaluates 24 items which assess the ability of walking, running and jumping and 4 points ordinals scale (0 to 3) will be scored. A scoring key of 0 "does not initiate", 1 "initiates", 2 "partially completes", 3 "completed" is used. The score will be calculated into percentage. The possible score range is 0% to 100%. Higher percentage means better performance. An experienced physiotherapist in pediatric will instruct the children while video will be recorded.
The change in Pediatric balance scale (PBS) between pre-treatment and post-treatment | will be measured at two intervals; pre-treatment and immediately after treatment
  PBS is an adapted tool from berg balance scale to assess balance for children diagnosed with cerebral palsy (CP) with mild to moderate motor dysfunction. The scale is consisting of 14 items including siting, standing and change of position. 5 points ordinals scale (0 to 4) will be given. 0 is poorest and 4 is the best performance for each items. The participant will have 3 trials and the best of three trials will be considered for the scoring. Possible range of total score is 0 to 56.
The change in Six minutes' walk test (6MWT) between pre-treatment and post-treatment | will be measured at two intervals; pre-treatment and immediately after treatment
  6-miutes walk test will be performed to evaluate the endurance in 30-meter walkway with marked cones at each start and end point. It measures the distance a individual is able to walk over a total of six minutes in meter. The individual is allowed to self-pace and rest as needed as they traverse back an forth along a marked walkway.
The change in Ten meter walk test (10MWT) between pre-treatment and post-treatment | will be measured at two intervals; pre-treatment and immediately after treatment
  10MWT will be used to evaluate the gait speed in meter per second which is performed on 14- meter track with the use of walking aid if the child is using during ambulation. The participant will perform 3 trials and average time will be used for the speed in meter per second.
The change in Edinburg visual gait score (EVGS) between pre-treatment and post-treatment | will be measured at two intervals; pre-treatment and immediately after treatment
  EVGS assesses the gait quality and pattern by observation which can be used every day in practice in mobilizing children diagnosed with cerebral palsy when gait analysis instrument is not available. It's a tabulated system which can record 17 observational items for each lower extremity in which the selected items represent a feature of pathological gait of ambulatory children with cerebral palsy. Six anatomical level such as trunk , pelvis ,hip , knee and foot will be observed from recording video. Sagittal, coronal, and transverse planes will be assessed. The selected angle of the joint is calculated from data obtained during instrumented analysis gait of normal subject.

SECONDARY OUTCOMES:
The change in Gross motor function measure - Dimension D (GMFM D) between pre-treatment and post-treatment | will be measured at two intervals; pre-treatment and immediately after treatment
  it is consist of 13 items and will be used to evaluate the ability of standing. 4 points ordinals scale (0 to 3) will be scored. A scoring key of 0 "does not initiate", 1 "initiates", 2 "partially completes", 3 "completed" is used. The score will be calculated into percentage. The possible score range is 0% to 100%. Higher percentage means better performance. An experienced physiotherapist in pediatric will instruct the children while video will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Meeyoung Kim, PhD, Principal Investigator — University of Sharjah
Locations (1):
- University of Sharjah, University City, Emirate of Sharjah, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make individual parrticipant data and related data dictionaries available.
Supporting Information: Study Protocol, SAP
Time Frame: After 6 months and will become availbel for one year
Access Criteria: Not identified yet

REFERENCES:
- [Background] Ammann-Reiffer C, Bastiaenen CH, Meyer-Heim AD, van Hedel HJ. Effectiveness of robot-assisted gait training in children with cerebral palsy: a bicenter, pragmatic, randomized, cross-over trial (PeLoGAIT). BMC Pediatr. 2017 Mar 2;17(1):64. doi: 10.1186/s12887-017-0815-y. PMID 28253887
- [Background] Aurich-Schuler T, Warken B, Graser JV, Ulrich T, Borggraefe I, Heinen F, Meyer-Heim A, van Hedel HJ, Schroeder AS. Practical Recommendations for Robot-Assisted Treadmill Therapy (Lokomat) in Children with Cerebral Palsy: Indications, Goal Setting, and Clinical Implementation within the WHO-ICF Framework. Neuropediatrics. 2015 Aug;46(4):248-60. doi: 10.1055/s-0035-1550150. Epub 2015 May 26. PMID 26011438
- [Background] Hilderley AJ, Fehlings D, Lee GW, Wright FV. Comparison of a robotic-assisted gait training program with a program of functional gait training for children with cerebral palsy: design and methods of a two group randomized controlled cross-over trial. Springerplus. 2016 Oct 28;5(1):1886. doi: 10.1186/s40064-016-3535-0. eCollection 2016. PMID 27843743
- [Background] Jin LH, Yang SS, Choi JY, Sohn MK. The Effect of Robot-Assisted Gait Training on Locomotor Function and Functional Capability for Daily Activities in Children with Cerebral Palsy: A Single-Blinded, Randomized Cross-Over Trial. Brain Sci. 2020 Oct 30;10(11):801. doi: 10.3390/brainsci10110801. PMID 33143214
- [Background] Lefmann S, Russo R, Hillier S. The effectiveness of robotic-assisted gait training for paediatric gait disorders: systematic review. J Neuroeng Rehabil. 2017 Jan 5;14(1):1. doi: 10.1186/s12984-016-0214-x. PMID 28057016